CLINICAL TRIAL: NCT04805684
Title: Comparison of Two Different Lung Ultrasound Imaging Protocols in COVID -19 Pneumonia
Brief Title: Different Lung Ultrasound Imaging Protocols in COVID-19 Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2021
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Lung Ultrasound; Pneumonia; Covid19
MeSH Terms: conditions — Pneumonia; COVID-19

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator was unaware of patient information such as medical history, PCR (polymerase chain reaction) test result, laboratory measurements, and CT scan results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lung ultrasound 12 (Active Comparator): 12 zone lung ultrasonography protocol
  Interventions: Device: LUS Twelve area
- lung ultrasound 14 (Active Comparator): 14 zone lung ultrasonography protocol
  Interventions: Device: LUS Fourteen area

INTERVENTIONS:
Device: LUS Twelve area — Application of 12 areas (2 posterior, 2 lateral, and 2 anterior)lung ultrasonography protocol using the convex ultrasound probe (2-6 MHz)
  Arms: lung ultrasound 12
Device: LUS Fourteen area — Application of 14 areas (3 posterior, 2 lateral, and 2 anterior) lung ultrasonography protocol using the convex ultrasound probe (2-6 MHz)
  Arms: lung ultrasound 14

SUMMARY:
Lung ultrasonography (LUS) is also used in COVID 19 pneumonia for diagnostic and follow-up purposes.It has been demonstrated in different studies that it can be used for pathologies in pleural and lung tissue. LUS was applied by different researchers by dividing the lungs into 12 and 14 regions and the results were shared.

DETAILED DESCRIPTION:
In our study, we aimed to determine the correlation between lung findings of COVID 19 pneumonia and thoracic tomography with the results of LUS applied to different numbers (12 versus 14) of areas.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 85 years old
* Hospitalized in intensive care unit
* PCR (polymerase chain reaction) tested
* Thoracic CT applied

Exclusion Criteria:

* Previous lung operation
* Thoracic wall disorder
* Interstitial lung disease
* Patients who did not consent to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Correlation between Thoracic CT imaging results and LUS results | 6 hours
  Lung ultrasonography will be performed within 6 hours of the Thoracic CT.

SECONDARY OUTCOMES:
Characteristics of lesions | 6 hours
  Identifying the characteristics of the abnormal findings detected in Thoracic CT and LUS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No